CLINICAL TRIAL: NCT06002958
Title: Horyzons: Implementation and Integration in Clinical Practice
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reductions in available funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-0672
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Schizophreniform Disorders; Schizoaffective Disorder; Unspecified or Other Psychotic Disorders
Keywords: Digital Intervention; Social Media; Virtual Therapeutic Content; First Episode Psychosis; Implementation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- FEP Providers (No Intervention): Approximately 20 FEP providers (clinicians and peer support specialists) affiliated with first episode psychosis (FEP) clinics in North Carolina (OASIS, SHORE, Encompass, Eagle, AEGIS) will be recruited to share their perspectives of barriers and facilitators in implementing and integrating a digital intervention in clinical practice. They will be asked to complete a survey examining their perspective and beliefs at two time points (baseline, 9 months) as well as a qualitative interview based on the Consolidated Framework for Implementation Science at 9 months.
- FEP Clients (Experimental): Approximately 50 individuals experiencing FEP and receiving services from FEP clinics (OASIS, SHORE, Encompass, Eagle, AEGIS) or their step down care clinics (STEP and TIDES) will be recruited to participate in a digital platform, Horyzons, for 12 months (for individuals enrolled at the initial opening of the platform; at a minimum 3 months of engagement) as part of their clinical care. Participants will have access to and encouraged to use the therapeutic content as well as the moderated online community network during their time engaging with the platform. They will be asked to complete a small battery of measures at baseline, 6-months, 12 months for individuals enrolled at the initiation of the study, while those enrolled later due to rolling recruitment may experience less assessment visits due to closing of the platform at the end of August 2024.
  Interventions: Device: Horyzons USA

INTERVENTIONS:
Device: Horyzons USA — Client participants will be onboarded to the digital platform, including the different spaces and how to use the site. The site includes therapeutic content that is tailored to each individual and their current needs and experiences, including social anxiety, generalized anxiety, mood, and social functioning, and distress intolerance. Further, the platform includes a moderated social media function, where individuals and peer support specialists can post text, images, videos, and comments to connect and share their experiences. The site is monitored by graduated students and trained clinicians.
  Arms: FEP Clients

SUMMARY:
The primary aim of this trial is evaluating the barriers and enablers of implementing a digital intervention with both therapeutic content and social networking, Horyzons, as part of clinical care in first episode psychosis (FEP) clinics in North Carolina. Providers (clinicians and peers support specialists) will be recruited from FEP clinics to assess Horyzons implementation and integration within clinical care at three time points (baseline, 6 months, and 12 months). Further, individuals experiencing FEP between the ages of 16 and 35 receiving services from the FEP clinics will be recruited to engage with the platform over the course of 12 months. Due to the nature of the digital intervention being implemented across the state of North Carolina, all research visits will be conducted remotely via videoconferencing.

DETAILED DESCRIPTION:
Purpose: The primary objective is to assess the barriers and facilitators of integrating Horyzons, an evidence-based digital intervention, in outpatient mental health clinics in North Carolina that provide care to individuals with schizophrenia spectrum and other unspecified psychotic disorders. The primary aim is to evaluate and identify the unique barriers and facilitators in implementing Horyzons at each first episode psychosis (FEP) clinic as part of standard care and distinct implementation strategies. The secondary and tertiary aims are to evaluate client engagement with Horyzons and attrition as part of clinical care and assess the change in clients' psychological measures across in addition to their use of state-funded services (e.g., emergency department and social services) across the 12-month intervention.

Participants: To assess the first aim, the investigators will recruit 20 clinicians and/or peer specialists from the FEP clinics. To assess the first and second aim, the investigators will recruit 50 individuals with FEP (i.e., first episode of a schizophrenia spectrum and other unspecified psychotic disorders).

Procedures (methods): Service provider participants will be recruited over a 4-6 week period at their respective clinics. They will be asked to complete an adapted measure, the Cancer Prevention and Control Research Network (CPCRN) Federally Qualified Health Center (FQHC) Survey, assessing clinical readiness, leadership, acceptance, adoption, and perspective on evidence-based practices. Service providers will then participate in implementing and integrating Horyzons within clinical practice including preferred implementation strategy that is distinct for each clinic (e.g., Horyzons training, access to the platform by clinicians, ongoing technical support, attendance and update at monthly team meetings, etc.). Service providers will meet with research staff at approximately the 6-month timepoint (+/- 4 weeks) to complete the CPCRN FQHC Survey then upon completion of the effectiveness trial with clients, service providers will complete this measure once again in addition to participating in a qualitative interview based on the Consolidated Framework for Implementation Research (CFIR) around their experience with integrating the platform and identification of barriers and facilitators to Horyzons' implementation. Service providers will be compensated for the completion feedback, including the questionnaire and qualitative interviews.

Client participants will be recruited over a 16- to 20-week period at their respective clinic. Participants will participate in a baseline visit to provide informed consent and complete a brief battery of measures (Demographics and Characteristics, University of California, Los Angeles (UCLA) Loneliness Scale, MOS Social Supports Survey). Participants will then meet with a research assistant, peer support specialist, or clinician to be given guidance and instruction for using the site (i.e., Horyzons onboarding). Clients will then engage in the platform, where site usage information as well as experience will be collected from participants through the Horyzons platform. Site usage (e.g., number of posts/comments made on the online platform, number and type of 'Journeys' or 'Tracks', self-guided therapeutic content, completed during time on the platform) will automatically be collected via the platform. Participants will have access and engage in this platform for approximately 12 months, depending on when recruited into trial. During this 12 month engagement period with the platform, client participants will meet with research staff at their midway point to complete the brief battery of measures assessing loneliness and social support and feedback on Horyzons. Upon completion of their engagement with the platform, client participants will additionally participate two additional research visits to complete the battery of measures at 12-months and at a 3-month follow-up. research visits to complete the battery of measures at 12-months and at a 3-month follow-up. As Horyzons involves therapeutic content and is designed to improve psychological outcomes, such as loneliness and social support, this platform is considered part of clinical care provided to individuals by their respective clinic. For this reason, participants will not be compensated for their usage and engagement with the platform, but rather, they will receive compensation for completion of assessment batteries at baseline, midway, final, and follow-up research study visits.

Horyzons will be monitored daily (two hours per weekday and one hour per weekend day) by trained peer support specialists, master's level clinicians, and/or graduate students with relevant clinical/research experience with individuals with psychosis. Drs. David Penn and Kelsey Ludwig, who are clinical psychologists, lead weekly supervision calls to ensure appropriate care and support of clients involved in the trial, to discuss case conceptualization and suggestions for engaging clients in the platform.

ELIGIBILITY:
CLIENT PARTICIPANTS

Inclusion Criteria:

* Clients must be between the ages of 16 and 35
* Clients must have a diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, or Unspecified Schizophrenia Spectrum or Other Psychotic disorder
* Clients must be receiving services at one of the five FEP clinics in North Carolina (OASIS, Encompass, Eagle, SHORE, or AEGIS) or one of their stepdown outpatient clinics (STEP and TIDES)
* Client not having any active thoughts of harming self in the month prior to enrollment
* Clients must not have been hospitalized for psychiatric reasons in the three months before enrollment
* Clients must actively be engaging with medication management through their clinic
* Clients must have access to the internet through a phone, tablet, or computer

Exclusion Criteria:

* Clients who do not speak English will not be considered for enrollment
* Adult client with legal guardians where one or both the individual and legal guardian do not provide consent for the individual to participate

PROVIDER PARTICIPANTS

Inclusion Criteria:

* Provider &/or PSS must be 18 years or older
* Provider &/or PSS must be currently serving clients within their FEP clinic
* Provider &/or PSS must be able to speak and read English

Exclusion Criteria:

* Provider &/or PSS under the age of 18
* Provider &/or PSS not currently serving clients in their FEP clinic
* Provider &/or PSS not able to speak or understand English

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Diana Perkins, MD, MPH, Principal Investigator — Univeristy of North Carolina, School of Medicine; Felice Reddy, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication and provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Requesting investigator has appropriate approval (see above) and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- FEP Providers: FEP providers (clinicians and peer support specialists) affiliated with first episode psychosis (FEP) clinics in North Carolina (OASIS, SHORE, Encompass, Eagle, AEGIS) will be recruited to share their perspectives of barriers and facilitators in implementing and integrating a digital intervention in clinical practice. They will be asked to complete a survey examining their perspective and beliefs at two time points (baseline, post-treatment) as well as a qualitative interview based on the Consolidated Framework for Implementation Science at the end of the trial.
- FEP Clients: Individuals experiencing FEP and receiving services from FEP clinics (OASIS, SHORE, Encompass, Eagle, AEGIS) or their step down care clinics (STEP and TIDES) will be recruited to participate in a digital platform, Horyzons, for 12 months (for individuals enrolled at the initial opening of the platform; at a minimum 3 months of engagement) as part of their clinical care. Participants will have access to and encouraged to use the therapeutic content as well as the moderated online community network during their time engaging with the platform. They will be asked to complete a small battery of measures at baseline, mid-treatment, post-treatment for individuals enrolled at the initiation of the study, while those enrolled later due to rolling recruitment may experience less assessment visits due to closing of the platform at the end of August 2024.
  Horyzons USA: Client participants will be onboarded to the digital platform, including the different spaces and how to use the site. The site includes therapeutic content that is tailored to each individual and their current needs and experiences, including social anxiety, generalized anxiety, mood, and social functioning, and distress intolerance. Further, the platform includes a moderated social media function, where individuals and peer support specialists can post text, images, videos, and comments to connect and share their experiences. The site is monitored by graduated students and trained clinicians.
Period: Overall Study
Arm/Group | FEP Providers | FEP Clients
Started | 20 | 32
Completed | 20 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FEP Providers | FEP Clients | Total
Number analyzed (Participants) | 20 | 32 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.75 (11.00) | 23.66 (4.44) | 29.08 (10.25)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 24 | 28
  Female | 14 | 8 | 22
  Non-Binary | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 20 | 29 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 11 | 12
  White | 18 | 15 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 32 | 52

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Summaries of Provider and Peer Support Specialists (PSSs) Participant Feedback in Post-Treatment Interview
Description: This qualitative data will be collected post-treatment from providers and PSSs. Individual interviews will discuss the utility and usage of Horyzons within their clinical care in addition to barriers and facilitators on numerous levels (individual, inner setting, and outer setting) of its implementation within their clinic. Feedback will be analyzed using grounded theory and summarized to include common themes regarding implementation, barriers, and enablers within the clinical setting and ideas for future implementation.
Time Frame: Up to 9 months
Population: This measure only applied to FEP Providers; therefore, data were not collected for FEP Clients.
Measure: Count of Participants; unit: Participants
Arm/Group | FEP Providers | FEP Clients
Number analyzed (Participants) | 20 | 0
Participants
  Viewed Horyzons as a way to combat loneliness and a safe space to socially engage with peers | 12 |
  Flexible/accessible resource that can be used anywhere and anytime | 10 |
  Therapy content that appealed to clients (e.g., psychoed and mindfulness exercises) | 10 |
  Platform lacks a true mobile app experience with notifications and updated design | 7 |
  Staff turnover and significant demands on clinicians' time made prioritizing Horyzons challenging | 10 |
  Lacked team integration; often viewed peer support and/or Horyzons as 'separate' | 9 |

2. Primary Outcome: Quantitative Summaries of Provider and PSS Participant Experience in Post-Treatment Feedback
Description: Quantitative data will be collected from providers and peer support specialists (PSSs) at baseline and post-treatment using a structured survey informed by the Consolidated Framework for Implementation Research (CFIR). The survey consists of Likert-style items rated from 1 = "strongly disagree" to 5 = "strongly agree" that capture perceived barriers and facilitators to implementing Horyzons in clinical practice (e.g., "People in our clinic actively seek new ways to improve how we do things").
  Items correspond to four subscales based on the CFIR framework: inner setting, outer setting, individual, and process. Subscale scores are calculated by averaging the items within each domain, after reverse scoring when appropriate. Each subscale ranges from 1 to 5, with higher scores indicating more positive perceptions of implementation support for Horyzons (i.e., better outcomes). Descriptive statistics (mean and standard deviation) are reported for each subscale.
Time Frame: Up to 9 months
Population: This measure only applied to FEP Providers; therefore, data were not collected for FEP Clients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Providers | FEP Clients
Number analyzed (Participants) | 20 | 0
score on a scale
  Inner (baseline) | 3.73 (0.43) |
  Inner (post-treatment) | 3.62 (0.19) |
  Outer (baseline) | 3.83 (0.70) |
  Outer (post-treatment) | 3.84 (0.54) |
  Individual (baseline) | 4.21 (0.48) |
  Individual (post-treatment) | 4.03 (0.48) |
  Process (baseline) | 3.77 (0.62) |
  Process (post-treatment) | 3.78 (0.49) |
Statistical Analysis 1: Comparison: FEP Providers; Test type: Other; Cohen's d = -0.29, 95% CI 2-sided [-0.815 to 0.255] — Inner
Statistical Analysis 2: Comparison: FEP Providers; Test type: Other; Cohen's d = 0.02, 95% CI 2-sided [-0.503 to 0.545] — Outer
Statistical Analysis 3: Comparison: FEP Providers; Test type: Other; Cohen's d = -0.32, 95% CI 2-sided [-0.850 to 0.225] — Individual
Statistical Analysis 4: Comparison: FEP Providers; Test type: Other; Cohen's d = 0.01, 95% CI 2-sided [-0.850 to 0.534] — Process

3. Secondary Outcome: Mean Change in UCLA Loneliness Scale Score
Description: The UCLA Loneliness scale is a 20-item scale. Answers are on a 4-point scale with options "I often feel this way," "I sometimes feel this way," "I rarely feel this way," and "I never feel this way." Possible scores range from 20 to 80. Higher scores reflect worse outcomes (greater feelings of loneliness). The UCLA Loneliness Scale is a part of the PhenX Toolkit.
Time Frame: Up to 9 months
Population: This measure only applied to FEP Clients; therefore, data were not collected for FEP Providers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Providers | FEP Clients
Number analyzed (Participants) | 0 | 32
score on a scale
  Baseline to Mid-treatment |  | -0.101 (9.61)
  Baseline to Post-treatment |  | -0.182 (9.61)

4. Secondary Outcome: Mean Change in Medical Outcomes Study (MOS) Social Support Survey - Total Score
Description: The MOS Social Support Survey is a 19-item scale. Answers are on a 5-point scale with options "none of the time", "a little of the time", "some of the time", "most of the time", and "all of the time". Possible scores range from 19 to 95. Higher scores reflect higher feelings of social support (more perceived social support). The mean change from baseline to mid-treatment and baseline to post-treatment will be averaged to get the overall mean for each timepoint. The MOS Social Support Survey is a part of the PhenX Toolkit.
Time Frame: Up to 9 months
Population: This measure only applied to FEP Clients; therefore, data were not collected for FEP Providers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Providers | FEP Clients
Number analyzed (Participants) | 0 | 32
score on a scale
  Baseline to Mid-treatment |  | -0.005 (11.66)
  Baseline to Post-treatment |  | 0.155 (11.66)

5. Secondary Outcome: Quantitative Summaries of Participant Experience in Post-Treatment Feedback
Description: This quantitative data will be collected post-treatment from clients. Feedback forms will prompt participants to answer questions regarding their experience with the platform on a scale of 1 to 5, with total scores ranging from 11-55 and higher scores reflecting a more positive experience.
Time Frame: Up to 9 months
Population: This measure only applied to FEP Clients; therefore, data were not collected for FEP Providers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Providers | FEP Clients
Number analyzed (Participants) | 0 | 32
score on a scale |  | 41.56 (7.50)

6. Other Pre Specified Outcome: Change in Use of Emergency and Social Services
Description: Collection of use of emergency and social services pre-initiation and post-initiation of Horyzons will be assessed to determine change in use of such services.
Time Frame: Baseline, up to Month 9
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Engagement With the Horyzons Platform and Attrition Over Time
Description: Changes in engagement with Horyzons will be passively collected for client participants via the platform. Data evaluated will include number of logins, number of journeys, tracks, and activities completed, and number engagements on the community page.
Time Frame: Baseline, up to Month 9
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, a total of approximately 9 months.
Arm/Group | FEP Providers | FEP Clients
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/32
Other Adverse Events (participants affected / at risk) | 0/20 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FEP Providers (N=20) | FEP Clients (N=32)
Inpatient Hospitalization due to Non-Adherence to Medication (Psychiatric disorders) | 0 (0) | 1 (1)
Inpatient Hospitalization due to Change in Medication Dosage (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT06002958/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT06002958/ICF_000.pdf